CLINICAL TRIAL: NCT02342990
Title: Telerehabilitation of Working Memory in Children With Periventricular Leukomalacia and Bilateral Cerebral Palsy, a Neuropsychological and Electrophysiological (High-density EEG) Study
Brief Title: Telerehabilitation of Working Memory in Children With Periventricular Leukomalacia and Bilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: University of Pisa (Other); University of Milan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC1/13-15_1.4
Record Dates: First submitted 2015-01-10; First posted 2015-01-21 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Periventricular Leukomalacia
Keywords: working memory training; home-based training; periventricular leukomalacia; bilateral cerebral palsy; neuropsychological profile; high density EEG; slow waves activities
MeSH Terms: conditions — Leukomalacia, Periventricular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cluster B (Experimental): After the first neuropsychological assessment (T1), children will start CogMed working memory training. Children will be retested (T2) about six or seven weeks later.
  Interventions: Other: Cluster B CogMed: an home-based and computer-based solution to improve working memory deficit
- Cluster A (Other): After the first neuropsychological assessment (T1), children will not start any training. Children will be retested (T2) about six or seven weeks later and will start CogMed working memory training. The group will be again retest (T3) after six or seven weeks after ended training.
  Interventions: Other: Cluster B CogMed: an home-based and computer-based solution to improve working memory deficit; Other: Cluster A No training. Delay start of CogMed

INTERVENTIONS:
Other: Cluster B CogMed: an home-based and computer-based solution to improve working memory deficit — CogMed: an home-based and computer-based solution to improve working memory deficit
Other: Cluster A No training. Delay start of CogMed — No training will be provided after T1 time point. Cluster A will start the CogMed training after the assessment at the T2 time point
  Arms: Cluster A

SUMMARY:
Periventricular Leukomalacia (PVL) is a white matter lesion surrounding the lateral ventricles of the brain occurring in the prenatal period, associated with a disorder of movement and posture, known as bilateral cerebral palsy. Children with PVL and bilateral cerebral palsy have spared verbal abilities, as measured by verbal Intelligence Quotient (verbal IQ) tests, while non-verbal intelligence and especially visuo-perceptual and visuo-spatial abilities are impaired. In addition some studies underline the impact of PVL also on executive function, especially in terms of working memory and in the ability to inhibit distraction.

Working Memory is the ability to retain and manipulate information for brief periods of time. It is important in several complex cognitive functions, such as academic learning and in planning and organizing daily life activities. School-based activities, indeed, such as math and reading depend on a student's ability to pay attention to several instructions or information and to hold and integrate them in their mind.

Recent behavioural and neurofunctional studies describes the effect of an evidence-based and computer-based training on working memory, the Cogmed Working MemoryTraining. Functional MRI show increase in parietal and prefrontal activity after this training, while the behavioural data demonstrate the generalization of this effect also on cognitive functions not directly trained, as attention, inhibition, learning and non-verbal reasoning. Cogmed Working MemoryTraining (RoboMemo®, CogMed-Cognitive Medical Systems, Stockholm, Sweden) is an online treatment comprising a number of visuo-spatial and verbal exercises that vary automatically depending on the individual child's performance in any given task. The training period is intensive and includes 25 home session for five weeks, 30-45 minutes each day. A Cogmed-trained coach monitors training progress and participants' commitment daily.

Only one ongoing study has used the CogMed training in children with cerebral palsy, but without investigating the correlation between behavioural findings with neurofunctional data.

The aim of this study is to analyze the effect of the working memory training with CogMed on trained and not directly trained cognitive abilities and on the changes in cortical electrophysiological reorganization during the sleep after training. The sleep analysis will be focused in particular on the slow waves activity [frequency range of 1-4.5 Hz] and on the sleep spindle [frequency range of 12-14Hz], which reflect the depth of sleep and are related to memory processes, learning and brain plasticity.

The results of this project will shed light on the mechanisms of neuroplasticity, by enhancing knowledge on the neuropsychological effects of a specific working memory training and on the neurophysiological underpinnings of these behavioural effects in a clinical population of children with congenital brain lesions, as PVL.

DETAILED DESCRIPTION:
The procedures implemented to register patients data will include the following steps:

* The quality assurance plan will provide: - to verify that all clinical fields, necessary to include and select patients, are available in the registry (e.g. type of cerebral palsy; MRI documentation, age); - to monitor that patients' contact information are available as well as testing materials and software; - to set team meetings to uniform recruitment procedure, data collection and registration.
* Data checks will be conducted by two or more researches from the team;
* Source data verification: both paper and electronic case report forms will be used and mutually checked.
* Data dictionary: Pre-post measures will be chosen by the team and described in a report form together with references and normative data.
* Procedure Standardization to address registry operations: Researches will co-work in patient recruitment and will attribute an identification number to each patient enrolled according to the inclusion and exclusion criteria evaluated by the neuropsychiatric team and described below. All researchers will be trained to register data in an internal database and to note the presence of adverse events. The researcher providing the training will assure comprehension and subscription of the written consent. Consent form will be discussed by the team in order to provide explicit and clear instructions on the training protocol to parents and patients.
* Calculation of sample size: Sample size, to specify the number of participants necessary to demonstrate the training effect, will be calculated from the training effect size between the Start index and the Max index provided by CogMed training. Based on a previous pilot study in our institute (effect size =.54) and on findings by Lundqvist and collaborators (2010) (effect size=.95), the effect size estimates for this study will be .60 and the sample size 20 children.
* Design: A stepped randomized clinical trial design will be chose to split the participants in two groups, matching for age and sex, in order to control test-retest effects. Both groups will receive neuropsychological and electrophysiological assessments at the same initial time point (T1). One group (Cluster B) will be start Cogmed training at home immediately after T1, while the second group (Cluster A) will start the training in the following time point (T2). When the training will be completed, both groups will be retested with neuropsychological and electrophysiological assessments (T2). After this time point, the Cluster A will start Cogmed training and will be re-tested with the same neuropsychological and the electrophysiological assessments at the finally time points (T3).
* The following time points will be provided:

Initial time point (T1) will correspond to pre-training assessment for both Clusters; Second time point (T2) will be provided after 6 or 7 weeks from T1 and will coincide with post-training assessment for the Cluster B and an other pre-training assessment for the Cluster A; Finally time point (T3), after 6 or 7 weeks from T2, will constitute the post-training assessment for Cluster A.

* Intervention program: Cogmed Working MemoryTraining (RoboMemo®, CogMed-Cognitive Medical Systems, Stockholm, Sweden) is an online treatment comprising a number of visuo-spatial and verbal exercises that vary automatically depending on the individual child's performance in any given task. The training period is intensive and includes 25 home session for five weeks, 30-45 minutes each day. A Cogmed-trained coach monitors training progress and participants' commitment daily for all the training period, corresponding to time period T1-T2 for Cluster B and T2-T3 for Cluster A.
* Plan for Missing data: Unavailable or not interpretable (significantly out of range) pre-post training data (behavioural or neurophysiological) will be considered as missing. The patients who will not complete the training will be excluded from the analysis.
* Plan for Statistical analysis: Univariate and Multivariate statistical analysis will be performed to compare neuropsychological performance and electrophysiological patterns at the different time points . Correlational analysis will be also performed to study the association between neuropsychological and electrophysiological data.

ELIGIBILITY:
Inclusion Criteria:

* PVL documented at brain MRI performed after age 2 years
* level I to III at the Manual Ability Classification System (MACS)
* IIntelligence Quotient above 80 in either verbal or non-verbal domains, as assessed by Wechsler preschool and primary scale of intelligence (WPPSI-III), Wechsler intelligence scale of children (WISC-III or WISC-IV) in the last year prior to recruitment

Exclusion Criteria:

* absence of a psychiatric disorder diagnosis or sensory deficits that preclude testing
* absence of drug-resistant epilepsy

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Working Memory (assessed by CogMed improvement index) | 5 weeks
  Working Memory will be assessed by CogMed improvement index, calculated subtracting the Start Index (the mean of the three best successful trials on days 2 and 3) from the Max Index (the mean of the three best successful trials on the two best training days).

SECONDARY OUTCOMES:
cortical electrophysiological reorganization during the sleep (high density EEG (hdEEG) | 6 or 7 weeks
  the electrophysiological signals will be register by high density EEG (hdEEG) during around one hour of sleep. The changing in the slow waves activity [frequency range of 1-4.5 Hz] and in the sleep spindle [frequency range of 12-14Hz], strongly associated with memory and learning mechanisms, will be analyze.
Short-term visuospatial memory (measured by Memory for Design subtest included in the Memory and Learning domain at the NEPSY-II) | 6 or 7 weeks
  Visuospatial memory assessment will be measured by Memory for Design subtest included in the Memory and Learning domain at the NEPSY-II. This subtest requires recognizing some designs and recalling its position on a grid (comprising from 4 to 10 designs) after a previous learning phase, both in immediately and delayed (after about 15-25 minutes) conditions. A raw scores for both immediately and delay conditions will be calculated.
Visual Attention (Executive Function/Attention domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  Visual attention is a visual search subtest included in Executive Function/Attention domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated.
Auditory Attention (assessed by Auditory Attention and Response Set subtest) | 6 or 7 weeks
  sustained auditory attention and the ability to shift and maintain new and complex set of rules, involving the inhibition of previously learned responses, will be assessed by Auditory Attention and Response Set subtest, included in Executive Function/Attention domain at the Developmental Neuropsychological battery (NEPSY-II). Raw scores will be calculated.
Inhibition (assessed by Inhibition subtests included in Executive Function/Attention domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  the ability to inhibit automatic responses in favour of novel responses and to switch between response types will be assessed by Inhibition subtests included in Executive Function/Attention domain at the Developmental Neuropsychological battery (NEPSY-II). Raw scores for accuracy and response time will be calculated.
phonological processing (assessed by Phonological processing subtest included in Executive Function/Attention domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  phonemic awareness and verbal working memory will be assessed by Phonological processing subtest included in Executive Function/Attention domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated.
visuo-graphical skills (assessed by Design Copy subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  the ability to copy complex geometric figures will be assessed by Design Copy subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated
visuo-constructional skills (evaluated by Block Construction subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  the ability to copy two-dimensional block models in three-dimensional representations with blocks will be evaluated by Block Construction subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated.
rotate mental representation (assessed by Geometric Puzzle subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  the ability to recognize rotated geometric shapes placed on a grid from a series of distractors will be assessed by Geometric Puzzle subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated
visuo-spatial skills (evaluated by Route Finding subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  the ability to identify the correct path leading to a house on a schematic map will be evaluated by Route Finding subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated.
visuo-perceptual skills (assessed by Arrows subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  visuo-perceptual abilities will be assessed by Arrows subtest included in the Visuospatial processing domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated.
Finger Tapping (assessed by Finger Tapping subtest included in the Sensorimotor skills domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  the ability to imitate a series of finger movements with the dominant and non-dominant hand will be assessed by Finger Tapping subtest included in the Sensorimotor skills domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated.
Imitating hand positions ( evaluated by Imitating hand position subtest included in the Sensorimotor skills domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  the ability to imitate hand and finger positions will be evaluated by Imitating hand position subtest included in the Sensorimotor skills domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated.
Visuo-motor Precision (assessed by Visuomotor Precision subtest included in Sensorimotor skills domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  visuo-motor control will be assessed by Visuomotor Precision subtest included in Sensorimotor skills domain at the Developmental Neuropsychological battery (NEPSY-II). Raw scores for accuracy and speed will be calculated.
Manual Motor Sequences (evaluated by Manual Motor Sequences included in the Sensorimotor skills domain at the Developmental Neuropsychological battery (NEPSY-II) | 6 or 7 weeks
  the ability to imitate and planning hand movements will be evaluated by Manual Motor Sequences included in the Sensorimotor skills domain at the Developmental Neuropsychological battery (NEPSY-II). Raw score will be calculated.

OTHER OUTCOMES:
child's behavior (CogMed parent rating scale questionnaire) | 6 or 7 weeks
  CogMed parent rating scale questionnaire will be filled out by the parents for monitoring child's behavior before and after training period. The questionnaire collect quantitative data on changes in the child's behaviour measuring raw scores for the follows behavioural area: attention, hyperactive and impulsive. This questionnaire will be filled only by parents of school-age children, as provided by CogMed.
Mathematic abilities (assess by one of the most widely used Italian mathematic battery, Test di valutazione delle ablitià di calcolo (AC-MT) | 6 or 7 weeks
  Mathematic abilities will be assess by one of the most widely used Italian mathematic battery, Test di valutazione delle ablitià di calcolo (AC-MT). For this project will be administered only the second part of battery, called individual condition, which include different subtests to assess mental and written calculation, arithmetic facts and numerical knowledge. Standard score will be provided.
Verbal Working memory span (assessed by the Following Instructions test provided by the CogMed program) | 3 weeks
  The Verbal working memory span will be assessed by the Following Instructions test provided by the CogMed program. In the Following Instruction test the child listen to a set of instructions and then click on or drag objects seen on the screen in a specific order. Test scores are expressed in span scores.
Visuospatial working memory span (assessed by the Working Memory test provided by the CogMed program) | 3 weeks
  The visuospatial working memory span will be assessed by the Working Memory test provided by the CogMed program. The Working Memory test is an exercise where the child have to identify the different shape from a set of three and remember its location. Test scores are expressed in span scores.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Gioni, MD, Study Chair — IRCCS-Stella Maris, Calambrone, Italy
Locations (1):
- IRCCS Stella Maris Foundation, Calambrone, Pisa, Italy